CLINICAL TRIAL: NCT04133922
Title: Effect of GLP-1 on Microvascular Insulin Responses in Type 1 Diabetes
Acronym: KML001
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: the study drug could not be obtained
Sponsor: University of Virginia (Other)
Collaborators: American Diabetes Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Zhenqi Liu, Deparment of Medicine, Chief of Div. Endocrinology, University of Virginia, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21590; 5R01DK102359-03 (NIH)
Record Dates: First submitted 2019-10-15; First posted 2019-10-21 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes; Insulin Sensitivity/Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Glucagon-Like Peptide 1; Insulin; Glucose; Water

STUDY DESIGN:
Intervention Model Description: Each subject is studied 3 times in randomized order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GLP-1 (Active Comparator): GLP-1 infusion 1.2 pmol/kg/min for 150 min
  Interventions: Drug: GLP-1
- GLP-1 + Insulin clamp (Active Comparator): GLP-1 infusion 1.2 pmol/kg/min for 150 min and insulin 1 mU/kg/min + Dextrose 20% at variable rate to maintain euglycemia for 120 min
  Interventions: Drug: GLP-1; Drug: Insulin; Drug: Dextrose 20 % in Water
- Saline + Insulin clamp (Active Comparator): Saline infusion at 30 ml/hr for 150 min and insulin 1 mU/kg/min + Dextrose 20% at variable rate to maintain euglycemia for 120 min.
  Interventions: Drug: Insulin; Drug: Dextrose 20 % in Water

INTERVENTIONS:
Drug: GLP-1 — glucagon-like peptide 1
  Arms: GLP-1; GLP-1 + Insulin clamp
Drug: Insulin — we are using to replace basal insulin and to raise insulin concentrations during the insulin clamp
  Arms: GLP-1 + Insulin clamp; Saline + Insulin clamp
Drug: Dextrose 20 % in Water — We are using Dextrose to maintain Euglycemia during the insulin clamp
  Arms: GLP-1 + Insulin clamp; Saline + Insulin clamp

SUMMARY:
GLP-1 increases skeletal and cardiac microvascular perfusion and improves insulin's microvascular responses in human subjects with T1DM, leading to improved metabolic insulin responses, endothelial function, and increased muscle oxygenation

DETAILED DESCRIPTION:
The proposed study will determine the effect of GLP-1 infusion on microvascular perfusion and microvascular insulin responses in both skeletal and cardiac muscle microvasculature in humans with T1DM. The investigators will study 20 participants with T1DM using a state-of-the-art technology, contrast enhanced ultrasound (CEU), to assess whether GLP-1 augments skeletal and cardiac microvascular blood flow (MBF) as a representation of microvascular perfusion, flow-mediated dilation (FMD) as a measurement of endothelial function, and augmentation index (AI) and pulse wave velocity (PWV) as surrogates for large vessel compliance. The investigators will use the combined CEU and euglycemic-hyperinsulinemic clamp approach to determine if microvascular and metabolic IR improves as a result.

ELIGIBILITY:
Inclusion Criteria:

1. History of type 1 diabetes, duration > 1 year
2. Age 18-40 years
3. HbA1c < 8.5%
4. BMI >/=18, <30 kg/m2
5. Using insulin for diabetes treatment only
6. On stable regimen of non-diabetic medications for the last 6 months, excluding oral contraceptives (OCP)
7. All screening labs within normal limits or not clinical significant

Exclusion Criteria:

1) Pregnancy or currently breastfeeding 2) Smoking history within 6 months 3) History of microvascular (microalbuminuria, retinopathy, neuropathy) or macrovascular diabetes complications (coronary artery disease, stroke, peripheral vascular disease) 4) Taking vasoactive medications (i.e. calcium channel blockers, angiotensin-converting enzyme or renin inhibitors, angiotensin-receptor blockers, nitrates, alpha-blockers) 5) OCP use within 3 months or 1 month if menses has subsequently occurred 6) Known hypersensitivity to perflutren (contained in Definity© contrast) 7) Screening O2 saturation<90% 8) Anemia (hemoglobin <12 g/dL in women, hemoglobin <13 g/dL in men) 9) Diabetic ketoacidosis (DKA) on presentation to screening visits or study admission days

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
change in microvascular blood volume between baseline and 2 hour insulin clamp | baseline and after 2 hour insulin clamp
  vascular measurement
change in insulin sensitivity between baseline and 2 hour insulin clamp | baseline and after 2 hour insulin clamp
  vascular measurement

SECONDARY OUTCOMES:
change in augmentation index between baseline and 2 hour insulin clamp | baseline and after 2 hour insulin clamp
  vascular measurement
change in flow-mediated dilation between baseline and 2 hour insulin clamp | baseline and after 2 hour insulin clamp
  vascular measurement
change in pulse wave velocity between baseline and 2 hour insulin clamp | baseline and after 2 hour insulin clamp
  vascular measurement

CONTACTS AND LOCATIONS:
Overall Officials: Zhenqi Liu, MD, Principal Investigator — Department of Endocrinology, University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Secrest AM, Becker DJ, Kelsey SF, Laporte RE, Orchard TJ. Cause-specific mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes. Diabetes. 2010 Dec;59(12):3216-22. doi: 10.2337/db10-0862. Epub 2010 Aug 25. PMID 20739685
- [Background] Krolewski AS, Kosinski EJ, Warram JH, Leland OS, Busick EJ, Asmal AC, Rand LI, Christlieb AR, Bradley RF, Kahn CR. Magnitude and determinants of coronary artery disease in juvenile-onset, insulin-dependent diabetes mellitus. Am J Cardiol. 1987 Apr 1;59(8):750-5. doi: 10.1016/0002-9149(87)91086-1. PMID 3825934
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263
- [Background] Soedamah-Muthu SS, Fuller JH, Mulnier HE, Raleigh VS, Lawrenson RA, Colhoun HM. High risk of cardiovascular disease in patients with type 1 diabetes in the U.K.: a cohort study using the general practice research database. Diabetes Care. 2006 Apr;29(4):798-804. doi: 10.2337/diacare.29.04.06.dc05-1433. PMID 16567818
- [Background] Peters SAE, Woodward M. Sex Differences in the Burden and Complications of Diabetes. Curr Diab Rep. 2018 Apr 18;18(6):33. doi: 10.1007/s11892-018-1005-5. PMID 29671082
- [Background] Huxley RR, Peters SA, Mishra GD, Woodward M. Risk of all-cause mortality and vascular events in women versus men with type 1 diabetes: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2015 Mar;3(3):198-206. doi: 10.1016/S2213-8587(14)70248-7. Epub 2015 Feb 6. PMID 25660575
- [Background] Di Carli MF, Afonso L, Campisi R, Ramappa P, Bianco-Batlles D, Grunberger G, Schelbert HR. Coronary vascular dysfunction in premenopausal women with diabetes mellitus. Am Heart J. 2002 Oct;144(4):711-8. PMID 12360169
- [Background] Mendelsohn ME, Karas RH. The protective effects of estrogen on the cardiovascular system. N Engl J Med. 1999 Jun 10;340(23):1801-11. doi: 10.1056/NEJM199906103402306. No abstract available. PMID 10362825
- [Background] Bjornstad P, Maahs DM, Duca LM, Pyle L, Rewers M, Johnson RJ, Snell-Bergeon JK. Estimated insulin sensitivity predicts incident micro- and macrovascular complications in adults with type 1 diabetes over 6 years: the coronary artery calcification in type 1 diabetes study. J Diabetes Complications. 2016 May-Jun;30(4):586-90. doi: 10.1016/j.jdiacomp.2016.02.011. Epub 2016 Feb 11. PMID 26936306
- [Background] Baron AD. Hemodynamic actions of insulin. Am J Physiol. 1994 Aug;267(2 Pt 1):E187-202. doi: 10.1152/ajpendo.1994.267.2.E187. PMID 8074198
- [Background] Millstein RJ, Pyle LL, Bergman BC, Eckel RH, Maahs DM, Rewers MJ, Schauer IE, Snell-Bergeon JK. Sex-specific differences in insulin resistance in type 1 diabetes: The CACTI cohort. J Diabetes Complications. 2018 Apr;32(4):418-423. doi: 10.1016/j.jdiacomp.2018.01.002. Epub 2018 Jan 10. PMID 29449137
- [Background] DeFronzo RA, Hendler R, Simonson D. Insulin resistance is a prominent feature of insulin-dependent diabetes. Diabetes. 1982 Sep;31(9):795-801. doi: 10.2337/diab.31.9.795. No abstract available. PMID 6761214
- [Background] Kaul K, Apostolopoulou M, Roden M. Insulin resistance in type 1 diabetes mellitus. Metabolism. 2015 Dec;64(12):1629-39. doi: 10.1016/j.metabol.2015.09.002. Epub 2015 Sep 11. PMID 26455399
- [Background] Priya G, Kalra S. A Review of Insulin Resistance in Type 1 Diabetes: Is There a Place for Adjunctive Metformin? Diabetes Ther. 2018 Feb;9(1):349-361. doi: 10.1007/s13300-017-0333-9. Epub 2017 Nov 14. PMID 29139080
- [Background] Gao F, Gao E, Yue TL, Ohlstein EH, Lopez BL, Christopher TA, Ma XL. Nitric oxide mediates the antiapoptotic effect of insulin in myocardial ischemia-reperfusion: the roles of PI3-kinase, Akt, and endothelial nitric oxide synthase phosphorylation. Circulation. 2002 Mar 26;105(12):1497-502. doi: 10.1161/01.cir.0000012529.00367.0f. PMID 11914261
- [Background] Clark MG. Impaired microvascular perfusion: a consequence of vascular dysfunction and a potential cause of insulin resistance in muscle. Am J Physiol Endocrinol Metab. 2008 Oct;295(4):E732-50. doi: 10.1152/ajpendo.90477.2008. Epub 2008 Jul 8. PMID 18612041
- [Background] Baron AD, Brechtel-Hook G, Johnson A, Cronin J, Leaming R, Steinberg HO. Effect of perfusion rate on the time course of insulin-mediated skeletal muscle glucose uptake. Am J Physiol. 1996 Dec;271(6 Pt 1):E1067-72. doi: 10.1152/ajpendo.1996.271.6.E1067. PMID 8997227
- [Background] Baron AD, Laakso M, Brechtel G, Edelman SV. Mechanism of insulin resistance in insulin-dependent diabetes mellitus: a major role for reduced skeletal muscle blood flow. J Clin Endocrinol Metab. 1991 Sep;73(3):637-43. doi: 10.1210/jcem-73-3-637. PMID 1874938
- [Background] Laakso M, Edelman SV, Brechtel G, Baron AD. Decreased effect of insulin to stimulate skeletal muscle blood flow in obese man. A novel mechanism for insulin resistance. J Clin Invest. 1990 Jun;85(6):1844-52. doi: 10.1172/JCI114644. PMID 2189893
- [Background] Barrett EJ, Wang H, Upchurch CT, Liu Z. Insulin regulates its own delivery to skeletal muscle by feed-forward actions on the vasculature. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E252-63. doi: 10.1152/ajpendo.00186.2011. Epub 2011 May 24. PMID 21610226
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Ratner R, Whitehouse F, Fineman MS, Strobel S, Shen L, Maggs DG, Kolterman OG, Weyer C. Adjunctive therapy with pramlintide lowers HbA1c without concomitant weight gain and increased risk of severe hypoglycemia in patients with type 1 diabetes approaching glycemic targets. Exp Clin Endocrinol Diabetes. 2005 Apr;113(4):199-204. doi: 10.1055/s-2005-837662. PMID 15891954
- [Background] Kim S, Jeong J, Jung HS, Kim B, Kim YE, Lim DS, Kim SD, Song YS. Anti-inflammatory Effect of Glucagon Like Peptide-1 Receptor Agonist, Exendin-4, through Modulation of IB1/JIP1 Expression and JNK Signaling in Stroke. Exp Neurobiol. 2017 Aug;26(4):227-239. doi: 10.5607/en.2017.26.4.227. Epub 2017 Aug 31. PMID 28912645
- [Background] Mazidi M, Karimi E, Rezaie P, Ferns GA. Treatment with GLP1 receptor agonists reduce serum CRP concentrations in patients with type 2 diabetes mellitus: A systematic review and meta-analysis of randomized controlled trials. J Diabetes Complications. 2017 Jul;31(7):1237-1242. doi: 10.1016/j.jdiacomp.2016.05.022. Epub 2016 May 30. PMID 28479155
- [Background] Dai Y, Mehta JL, Chen M. Glucagon-like peptide-1 receptor agonist liraglutide inhibits endothelin-1 in endothelial cell by repressing nuclear factor-kappa B activation. Cardiovasc Drugs Ther. 2013 Oct;27(5):371-80. doi: 10.1007/s10557-013-6463-z. PMID 23657563
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Nystrom T, Gutniak MK, Zhang Q, Zhang F, Holst JJ, Ahren B, Sjoholm A. Effects of glucagon-like peptide-1 on endothelial function in type 2 diabetes patients with stable coronary artery disease. Am J Physiol Endocrinol Metab. 2004 Dec;287(6):E1209-15. doi: 10.1152/ajpendo.00237.2004. Epub 2004 Sep 7. PMID 15353407
- [Background] Chai W, Zhang X, Barrett EJ, Liu Z. Glucagon-like peptide 1 recruits muscle microvasculature and improves insulin's metabolic action in the presence of insulin resistance. Diabetes. 2014 Aug;63(8):2788-99. doi: 10.2337/db13-1597. Epub 2014 Mar 21. PMID 24658303
- [Background] Chai W, Fu Z, Aylor KW, Barrett EJ, Liu Z. Liraglutide prevents microvascular insulin resistance and preserves muscle capillary density in high-fat diet-fed rats. Am J Physiol Endocrinol Metab. 2016 Sep 1;311(3):E640-8. doi: 10.1152/ajpendo.00205.2016. Epub 2016 Jul 19. PMID 27436611
- [Background] Basu A, Charkoudian N, Schrage W, Rizza RA, Basu R, Joyner MJ. Beneficial effects of GLP-1 on endothelial function in humans: dampening by glyburide but not by glimepiride. Am J Physiol Endocrinol Metab. 2007 Nov;293(5):E1289-95. doi: 10.1152/ajpendo.00373.2007. Epub 2007 Aug 21. PMID 17711996